CLINICAL TRIAL: NCT01423695
Title: Weekly Application of Trastuzumab and Paclitaxel in the Treatment of HER2-overexpressing Metastatic Breast Cancer
Brief Title: Weekly Paclitaxel and Trastuzumab in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: WiSP Wissenschaftlicher Service Pharma GmbH (Other)
Collaborators: Bristol-Myers Squibb (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WISP_RO78
Record Dates: First submitted 2011-08-25; First posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- paclitaxel/trastuzumab (Experimental): Single experimental arm in a phase II trial
  Interventions: Drug: paclitaxel plus trastuzumab

INTERVENTIONS:
Drug: paclitaxel plus trastuzumab — Weekly paclitaxel (90 mg/m² iv, 12 courses) plus weekly trastuzumab (4mg/kg body weight iv as loading dose, 2 mg/kg iv from week 2 onwards; continued until disease progression)

SUMMARY:
The 3 weekly combination of trastuzumab and paclitaxel has been approved for the treatment of advanced breast cancer based on a large pivotal study. However, mono and combination chemotherapy trials suggest that weekly paclitaxel has a better therapeutic index, especially in the palliative setting. The present trial examines the efficacy and safety of weekly paclitaxel over a limited duration combined with continued trastuzumab in HER2+ patients.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed metastatic breast cancer overexpressing HER2
* pretreatment with anthracycline in either the adjuvant or palliative setting.
* HER2 positivity was defined as 2+ or 3+ overexpression using the DAKO HercepTest, confirmed by fluorescence in-situ hybridization (FISH) if 2+.
* informed consent

Exclusion Criteria:

* more than 1 chemotherapy for advanced disease
* taxane or trastuzumab pretreatment
* brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status >1
* pregnancy or lactation, childbearing potential without reliable contraception
* clinically significant cardiac disease,
* neutrophils <1500/µl, platelets <75,000/µl
* total bilirubin and creatinine >1.5 × the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2001-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Patient follow-up on average for 15 months and up to a maximum of 51 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthias John, MD, Principal Investigator — Oncology Practice, Glauchau
Locations (1):
- Dr. Matthias John, Glauchau, Saxony, Germany